CLINICAL TRIAL: NCT06402305
Title: Lipid Profile and Ultrasound Findings in Patients With Pancreaticobiliary Diseases
Status: Recruiting | Type: Observational
Sponsor: Alaa Mohamed Mostafa (Other)
Responsible Party: Sponsor-Investigator, Alaa Mohamed Mostafa, Resident in Tropical Medicine and Gastroenterology Department Sohag University Hospital, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med-24-04-015MS
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Lipid Profile and Ultrasound Findings in Patients With Pancreaticobiliary Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: Cases
  Interventions: Diagnostic Test: Lipid profile
- group B: Controls
  Interventions: Diagnostic Test: Lipid profile

INTERVENTIONS:
Diagnostic Test: Lipid profile — Abdominal ultrasound and lipid profile will be done
  Other Names: Abdominal ultrasound

SUMMARY:
Gall stones happen is the most prevalent pathology affecting the biliary system due to its Physiological function of concentration of bile having a prevalence of 10%-15% and an incidence of 1.4% per year in the adult population of developed countries (Halldestam et al,. 2009). Women are more commonly affected by gall stone disease as compared to men (Attili et al,. 1995).

Multiple risk factors responsible for the Gall stone formation include modifiable factors such as lifestyle factors (reduced physical activity, rapid weight loss, fasting, and oral contraceptives (Di Ciaula et al,. 2013); dietary factors (high fat, high cholesterol, high refined carbohydrates, and low fiber ; metabolic syndrome (obesity, diabetes mellitus, dyslipidemia, and hyperinsulinemia (Cuevas et al., 2004).

Among all the above mentioned risk factors, serum lipids are considered to be the most important risk factor involved in the pathogenesis of Gall stone disease (Celika et al,. 2015). Hyperlipidemia is generally characterized by high serum levels of total cholesterol, triglycerides, low density lipoproteins (LDL-C), and low levels of high-density lipoprotein (HDL-C). Some studies have showed a significant association of hyperlipidemia with gall stones especially hypertriglyceridemia and increased LDL-C levels (Rao et al,. 2012).

Acute pancreatitis (AP) is an inflammatory condition of the pancreas that originates within the pancreatic acinar cells and causes pancreatic necrosis, systemic inflammatory response syndrome, and multiple organ failure (Crockett et al,. 2013). According to The revised Atlanta classification system from 2012 ,AP is diagnosed on the basis of two of three criteria-typically belt-like abdominal pain, an elevated serum lipase level three times above the normal threshold, and radiological imaging signs of pancreatitis (Parniczky et al,.2016).

Severe hypertriglyceridemia is a well-known cause of AP. Recent studies have suggested that elevated serum triglyceride and low high-density lipoprotein cholesterol (HDL-C) levels are associated with persistent organ failure in acute pancreatitis (Peng et al,. 2015). With the change of people's diet structure and lifestyle, the incidence and mortality of hypertriglyceridemic AP are increasing year by year and has surpassed alcohol as the second leading cause of AP (Carr et al,. 2016).

Chronic pancreatitis is a syndrome characterized by chronic progressive pancreatic inflammation, fibrosis, and scarring, resulting in damage to and loss of exocrine (acinar), endocrine (islet cells), and ductal cells(Majumder S,. 2016)

ELIGIBILITY:
Inclusion Criteria:

* Patients with age above 18 years
* Patients with confirmed diagnosis of gall stones ,acute calcular cholecystitis ,calcular obstructive jaundice ,biliary stricture ,acute and chronic pancreatitis

Exclusion Criteria:

* Patients with renal failure, hemolytic diseases (hereditary spherocytosis, sickle cell anemia on history and CBC film).
* Patients on antihyperlipidemic drugs .

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adiagnosis of gall stones ,acute calcular cholecystitis,calcular obstructive jaundice ,biliary stricture ,acute and chronic pancreatitis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-05-05 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
Lipid Profile and Ultrasound Findings in Patients with Pancreaticobiliary Diseases | 1 year
  * To evaluate the lipid profile and ultrasound findings in biliary diseases
  * To assess the lipid profile and ultrasound findings in pancreatic diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Attili AF, Carulli N, Roda E, Barbara B, Capocaccia L, Menotti A, Okoliksanyi L, Ricci G, Capocaccia R, Festi D, et al. Epidemiology of gallstone disease in Italy: prevalence data of the Multicenter Italian Study on Cholelithiasis (M.I.COL.). Am J Epidemiol. 1995 Jan 15;141(2):158-65. doi: 10.1093/oxfordjournals.aje.a117403. PMID 7817971
- [Background] Carr RA, Rejowski BJ, Cote GA, Pitt HA, Zyromski NJ. Systematic review of hypertriglyceridemia-induced acute pancreatitis: A more virulent etiology? Pancreatology. 2016 Jul-Aug;16(4):469-76. doi: 10.1016/j.pan.2016.02.011. Epub 2016 Mar 3. PMID 27012480
- [Background] Crockett SD, Wani S, Gardner TB, Falck-Ytter Y, Barkun AN; American Gastroenterological Association Institute Clinical Guidelines Committee. American Gastroenterological Association Institute Guideline on Initial Management of Acute Pancreatitis. Gastroenterology. 2018 Mar;154(4):1096-1101. doi: 10.1053/j.gastro.2018.01.032. Epub 2018 Feb 3. No abstract available. PMID 29409760
- [Background] Halldestam I, Kullman E, Borch K. Incidence of and potential risk factors for gallstone disease in a general population sample. Br J Surg. 2009 Nov;96(11):1315-22. doi: 10.1002/bjs.6687. PMID 19847878